CLINICAL TRIAL: NCT00694837
Title: Phase I/II Study for Patients With Newly Diagnosed Glioblastoma Testing Nelfinavir in Combination With Concomitant Temozolomide and Radiotherapy.
Brief Title: Study With Nelfinavir and Combined Radiochemotherapy for Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-09-04/07; EudraCT number 2008-001078-34
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Glioblastoma
Keywords: glioblastoma; nelfinavir; functional imaging; AKT pathway
MeSH Terms: conditions — Glioblastoma | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- B (Experimental)
  Interventions: Drug: nelfinavir

INTERVENTIONS:
Drug: nelfinavir — The start dose of nelfinavir in phase 1 is 1000mg BID. The maximum administered dose, if no DLT occurs, will be1250 mg BID (2500mg). Nelfinavir will be administered 1 week before start of the chemoradiotherapy until the last day of chemoradiotherapy.

SUMMARY:
The objectives of the trial are:

To assess safety, tolerability and activity of nelfinavir given neo-adjuvant and concomitant to chemoradiotherapy with temozolomide in patients with a newly diagnosed glioblastoma multiforme.

To describe the possible effect of nelfinavir on functional imaging To describe the activity of nelfinavir in vivo on blocking the AKT pathway.

DETAILED DESCRIPTION:
Glioblastoma multiforme is the most malignant and common, about 50%, variant of all primary brain tumours. The treatment strategies for this disease have not changed appreciably for many years consisting of a surgical intervention (biopsy or tumour resection) and post-operative local radiotherapy until several years ago. Combined chemoradiotherapy with temozolomide is at the moment the standard medical practice after results of the joint EORTC-NCIC phase III study randomizing between radiotherapy alone and combined chemoradiotherapy with temozolomide showed a significant improvement in 2-years survival from 8% to 24% for the combined treatment arm (Stupp 2005). Given the poor prognosis of these patients and the still poor treatment response, further therapeutic improvement will remain the most challenging topic for the future. The next step to further improve survival for this patient group would be the addition of biological modifying and/or antiangiogenic therapies. These strategies are motivated by the fact that glioblastomas often express very high levels of vascular endothelial growth factor which is a key mediator of blood vessel growth as high expression of EGFR, which upregulates the downstream PI3K-AKTpathway. (Fischer I, Carmeliet P, Koul D) One possible candidate is nelfinavir, a protease inhibitor interfering with Akt activity downstream of EGFR and upstream of VEGF. (Geng L, Gorski D, HLu B)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme at primary diagnosis
* Tumours which do enhance on pre-operative imaging
* Age >=18-65 years
* WHO performance status 0-2, RTOG- RPA class III-IV.
* No recent (< 3 months) severe cardiac disease (arrhythmia, congestive heart failure, infarction)
* Patient able to tolerate full course of radiotherapy
* No previous radiotherapy to the head and neck area.
* Prior neurosurgery within 6 weeks of treatment
* No previous irradiation of the brain.
* No previous chemotherapy
* No prior or concurrent medical condition which would make treatment difficult to complete. Medication with steroids is allowed.
* No use of terfenadine, astemizol, cisapride, sildenafil, lovastatin or simvastatin and other concurrent medication that is metabolized by the CYP3A4 isoenzyme and cannot be replaced with other equivalent medications for the period of the study: antiarrhythmics (amiodarone, quinidine), neuroleptics (pimozide), sedative/hypnotic agents (midazolam, triazolam), ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine), HMG-CoA reductase inhibitors (atorvastatin), rifampin, rifabutin, felodipine, nifedipine, and sildenafil or St. John's wort.
* Adequate haematological, renal and hepatic function
* No uncontrolled infectious disease, absence of known HIV infection, chronic hepatitis B or hepatitis C infection
* Absence of any medical condition, which could interfere with oral medication intake (e.g., frequent vomiting, partial bowel obstruction)
* All patients of reproductive potential (male and female) must use effective contraception for the whole duration of the treatment and until 6 months thereafter. Females must not be pregnant or lactating
* Willing and able to comply with the study prescriptions
* Written informed consent before patient registration

Exclusion Criteria:

The opposite from above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fase I: To determine the MTD of nelfinavir as an adjuvant in the radiochemotherapy treatment in primary glioblastoma patients. Fase 2: Progression free survival at 6 months | Fase 1: after treatment; fase 2: 6 months after treatment

SECONDARY OUTCOMES:
Fase 1/2: Incidence of acute toxicity; OS; Metabolic ratios of SUV of serial 18F-FDG: assessed by PET-CT.Fase 1:6-months PFS; Relative blood flow measurement by perfusion MRI. Fase 2: PFS at 12 months; Phosphorylation of AKT in tumour tissue. | fase 1: 6 months after treatment; fase 2: 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta Baumert, MD PhD, Principal Investigator — Maastricht Radiation Oncology
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Netherlands